CLINICAL TRIAL: NCT05443633
Title: Enhancing Language Function in Aphasia Using Behavioral Language Intervention
Brief Title: Enhancing Language Function in Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001134
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Aphasia, Acquired; Language Disorders; Primary Progressive Aphasia; Stroke, Cerebrovascular
MeSH Terms: conditions — Aphasia; Language Disorders; Aphasia, Primary Progressive; Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: individuals will be randomized to the active intervention or control group (standard care)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The subject codes will be used for blinding of the participants, care-providers, and assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active therapy group (Experimental): Participants will undergo individualized language treatment in which they will learn semantically- or phonologically based strategies to facilitate word finding difficulties, sentence formulation difficulties, or challenges in their narration and discourse. The level at which the treatment will be administered will depend on the participants' level of performance determined by the results of the language and cognitive testing done at baseline. Treatment will be administered twice a week for 10 weeks.
  Interventions: Behavioral: individualized speech-language training
- control group (Active Comparator): control group will undergo standard speech-language intervention
  Interventions: Behavioral: standard language intervention

INTERVENTIONS:
Behavioral: individualized speech-language training — Language treatment might include lexical, semantic, and interactive treatment. During treatment, patients may be trained to name words by attempting to self-cue lexical retrieval. The therapy moves incrementally through semantic cuing. The semantic treatment will be implemented using the methods described in (Edmonds et al., 2009, 2014).
  Other Names: active
  Arms: Active therapy group
Behavioral: standard language intervention — Participants will undergo standard speech-language naming therapy
  Other Names: control
  Arms: control group

SUMMARY:
Aphasia is an acquired impairment of language, that commonly results from damage to language areas in the brain (typically the left side of the brain). This impairment is seen in many aspects of language, including understanding, speaking, reading and writing. It is estimated that about 2 million individuals are currently living with aphasia in the United States. Further, about 200,000 Americans acquire aphasia every year (National Aphasia Association, 2020). Aphasia poses significant impact on the affected individuals and their families. Behavioral treatments that target language deficits have been shown to enhance overall communication skills and life satisfaction among individuals with aphasia. Although there is evidence that suggests that treatment is efficacious for individuals with aphasia, the extent of improvement long-term coupled with the neural patterns among those individuals are largely unknown. The current study aims to investigate the efficacy of language-based treatment and its corresponding neural patterns.

DETAILED DESCRIPTION:
The purpose of this study is to develop semantic-based treatment to address language deficits in individuals with acquired language disorders. We propose to develop an individually optimized semantic-based protocol for strategy implementation and word finding facilitation among individuals with language disorders.

Phase 1: Following screening, participants who fulfill the inclusion criteria and have consented to participate in the study will undergo baseline cognitive and language assessment, electroencephalography (EEG) recording and the magnetic resonance imaging (MRI) scan. Participants with language disorders will proceed to the following phases.

Phase 2: After baseline assessment, participants will undergo individualized language treatment in which they will learn semantically- or phonologically based strategies to facilitate word finding difficulties, sentence formulation, or challenges in their narration and discourse. The level at which the treatment will be administered will depend on the participants' level of performance determined by the results of the language and cognitive testing done at baseline. Treatment will be administered twice a week for 10 weeks.

Phase 3: Directly following treatment, patients will undergo cognitive and language assessment, EEG recording, and an MRI scan. This is done to test for short-term changes in behavioral abilities and neural patterns.

Phase 4: After 2 months after the treatment, participants will undergo cognitive and language assessment, EEG recording, and an MRI scan. This final phase of testing is done to test for long-term changes in behavioral abilities and neural responses.

ELIGIBILITY:
Inclusion Criteria:

1. Present with speech-language impairment (aphasia) caused by stroke or dementia
2. A medical diagnosis of primary progressive aphasia (PPA) by a neurologist or physician
3. Are native speakers of English
4. Present with no contraindications for MRI
5. Have adequate (normal or corrected to normal) vision and hearing

Exclusion Criteria:

1. Individuals diagnosed with mood, anxiety, psychotic or substance abuse disorders.
2. Individuals with highly magnetizable metallic implants, including certain dental work, may be excluded due to image quality in MRI.
3. Individuals with other neurological disorders besides the ones of interest for the study (e.g., epilepsy, Multiple Sclerosis, Parkinson's Disease)
4. Individuals with contraindications for MRI. This includes but is not limited to pacemakers, metallic cardiac pumps, valves, magnetic materials such as surgical clips, implanted electronic perfusion pumps, or any other condition that would preclude proximity to a strong magnetic field.
5. Individuals suffering from clinically significant claustrophobia
6. Severe systemic disease (e.g., renal failure)
7. Poor overall health
8. Individuals who are pregnant
9. Individuals with a history of epileptic activity in the past 12 months
10. Individuals with a personal or family history of epilepsy or other seizure disorders will not be included in the study.
11. Individuals who have had a brain surgery in the past
12. Individuals with implanted metallic skull plates or intracranial implants
13. Individuals with skin lesions or skull damage
14. Individuals who have a history of excessive use of alcohol or drugs
15. Individuals with premorbid psychiatric disease affecting communication
16. Individuals with severe non-linguistic cognitive disturbances impeding language therapy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline scores on the naming task | through study completion, an average of 1 year
  Mean change from baseline scores on the Boston Naming Test: Min score = 0; Max = 60; higher scores indicate better outcome
Mean change from baseline scores in aphasia severity | through study completion, an average of 1 year
  Mean change from baseline scores on the Western Aphasia Battery: Min score = 0; Max = 100; higher scores indicate better outcome
Mean change from baseline scores on the language probe task before and after each session | through study completion, an average of 1 year
  change on on the probe task from before the session; Min =0; Max = 100%; higher scores indicate better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Kielar, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No